CLINICAL TRIAL: NCT03083704
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Second Generation Andexanet Alfa Administered to Healthy Subjects
Brief Title: A Healthy Volunteer PK/PD, Safety and Tolerability Study of Second Generation Andexanet Alfa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-512
Record Dates: First submitted 2017-03-07; First posted 2017-03-20 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — PRT064445; apixaban; Rivaroxaban; enoxaparin sodium; edoxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Cohort 1 (Experimental)
  Interventions: Drug: Apixaban 5 MG; Biological: Andexanet alfa (Gen 1 Process 3)
- Cohort 2 (Experimental)
  Interventions: Drug: Rivaroxaban 20 MG; Biological: Andexanet alfa (Gen 1 Process 3)
- Cohort 3 (Experimental)
  Interventions: Biological: Andexanet alfa (Gen 1 Process 2); Drug: Apixaban 5 MG
- Cohort 4 (Experimental)
  Interventions: Drug: Apixaban 5 MG; Biological: Andexanet alfa (Gen 2)
- Cohort 5 (Experimental)
  Interventions: Drug: Rivaroxaban 20 MG; Biological: Andexanet alfa (Gen 2)
- Cohort 6 (Experimental)
  Interventions: Drug: Enoxaparin sodium; Biological: Andexanet alfa (Gen 2)
- Cohort 7 (Experimental)
  Interventions: Drug: Edoxaban 60 MG; Biological: Andexanet alfa (Gen 2)
- Cohort 8 (Experimental)
  Interventions: Biological: Andexanet alfa (Gen 2); Drug: Apixaban 10 MG
- Cohort 9 (Experimental)
  Interventions: Biological: Andexanet alfa (Gen 2); Drug: Rivaroxaban 10 MG
- Cohort 10 (Experimental)
  Interventions: Drug: Enoxaparin sodium; Biological: Andexanet alfa (Gen 2)
- Cohort 11 (Experimental)
  Interventions: Drug: Edoxaban 60 MG; Biological: Andexanet alfa (Gen 2)

INTERVENTIONS:
Biological: Andexanet alfa (Gen 1 Process 2) — factor Xa inhibitor antidote
  Arms: Cohort 3
Drug: Apixaban 5 MG — factor Xa inhibitor
  Arms: Cohort 1; Cohort 3; Cohort 4
Drug: Rivaroxaban 20 MG — factor Xa inhibitor
  Arms: Cohort 2; Cohort 5
Drug: Enoxaparin sodium — low molecular weight heparin
  Arms: Cohort 10; Cohort 6
Drug: Edoxaban 60 MG — factor Xa inhibitor
  Arms: Cohort 11; Cohort 7
Biological: Andexanet alfa (Gen 2) — factor Xa inhibitor antidote
  Arms: Cohort 10; Cohort 11; Cohort 4; Cohort 5; Cohort 6; Cohort 7; Cohort 8; Cohort 9
Biological: Andexanet alfa (Gen 1 Process 3) — factor Xa inhibitor antidote
  Arms: Cohort 1; Cohort 2
Drug: Apixaban 10 MG — factor Xa inhibitor
  Arms: Cohort 8
Drug: Rivaroxaban 10 MG — factor Xa inhibitor
  Arms: Cohort 9

SUMMARY:
This is a randomized, double-blind, study in healthy volunteers dosed to steady state with fXa inhibitors, designed to (1) demonstrate PK/PD comparability between andexanet manufactured by the Generation 1 and Generation 2 processes, (2) evaluate the degree to which the Generation 2 andexanet reverses fXa-inhibitor-induced anticoagulation in comparison to placebo, and (3) evaluate safety of Generation 2 andexanet.

ELIGIBILITY:
Inclusion Criteria:

1. Must be in reasonably good health as determined by the Investigator based on medical history, full physical examination (including blood pressure and pulse rate measurement), 12-lead ECG, and clinical laboratory tests. Subjects with well-controlled, chronic, stable conditions (e.g., controlled hypertension, non-insulin dependent diabetes, osteoarthritis, hypothyroidism) may be enrolled based on the clinical judgment of the Investigator and if approved by the Medical Monitor.
2. Must be between the ages of 18 and 75 years, inclusive, at the time of signing of the informed consent form (ICF).
3. Agrees to have any dietary or nutritional supplements reviewed by the Investigator and potentially be withheld during the study if advised by the Investigator. Standard multivitamin and mineral supplementation will be permitted.
4. Agrees to comply with the contraception and reproduction restrictions of the study:

   * Men whose sexual partner is of childbearing potential and/or who are not monogamous must be using two acceptable methods of contraception, at least one of which must be a barrier method (e.g., spermicidal gel plus condom), for the entire duration of the study and for at least 1 month following study-drug administration; and men must refrain from attempting to father a child or donating sperm in the 1 month following the study-drug administration. Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception;
   * Men who report surgical sterilization (e.g., bilateral vasectomy) must have had the procedure at least 6 months before study drug administration.
   * Surgical sterilization procedures should be supported with clinical documentation and noted in the Relevant Medical History/Current Medical Conditions section of the case report forms (CRFs).
   * Women of childbearing potential must be using two medically acceptable methods of contraception, at least one of which must be a barrier method (e.g., non-hormone containing intra-uterine device plus condom, spermicidal gel plus condom, diaphragm plus condom), from the time of Screening and for the duration of the study, through at least 1 month following study drug administration. NOTE: Oral and topical hormonal contraceptive use, as well as the use of hormone-containing intra-uterine devices, is not permitted due to their increased risk of thromboembolism. Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception; OR
   * Postmenopausal women must have had no regular menstrual bleeding for at least 1 year before initial dosing and either be over the age of 60 years or have an elevated plasma follicle-stimulating hormone (FSH) level (i.e., > 40 mIU/mL) at Screening; OR
   * Women who report surgical sterilization (i.e., hysterectomy, tubal ligation, and/or bilateral oophorectomy) must have had the procedure at least 6 months before study drug administration. Surgical sterilization procedures should be supported with clinical documentation and noted in the Relevant Medical History/Current Medical Conditions section of the CRF; AND
   * All female subjects must have a documented negative pregnancy test result at Screening and on Study Day 1.
5. Systolic blood pressure < 160 mmHg and diastolic blood pressure < 90 mmHg at Screening and Day 1.
6. The following laboratory values must be within the normal laboratory reference range within 28 days of Day 1: prothrombin time (PT), activated partial thromboplastin time (aPTT), and activated clotting time (ACT); hemoglobin, hematocrit, and platelet count.
7. The following laboratory values must be equal to or below 2 times the upper limit of normal (ULN) range within 28 days of Day 1: Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) and total bilirubin.
8. The Screening serum creatinine must be below 1.5 mg/dL within 28 days of Day 1.
9. Body mass index between 19-30 kg/m2, inclusive, and body weight at least 50 kg.
10. Agrees to abstain from alcohol consumption for the duration of the domicile period, and from the use of drugs of abuse for the duration of the study.
11. Able to read and give written informed consent and has signed a consent form approved by the Investigator's Institutional Review Board (IRB) or Independent Ethics Committee (IEC).

Exclusion Criteria:

1. Previous use of andexanet or previous participation in the current study.
2. History of abnormal bleeding, signs or symptoms of active bleeding, or risk factors for bleeding.
3. Has a stool specimen that was positive for occult blood within 6 months of study Screening or during the Screening Period.
4. Past or current medical history of thrombosis, any sign or symptom that suggests an increased risk of a systemic thrombotic condition or thrombotic event, or recent events that may increase risk of thrombosis.

   a. For example, subjects with a known or suspected hypercoagulable state, history of VTE, DVT, stroke, myocardial infarction [MI], cancer [other than non-melanoma skin cancer], atrial fibrillation, heart failure, cardiomyopathy, phlebitis, lower extremity edema, major surgery or trauma within 2 months of Study Day 1, airplane travel ≥ 2 hours during the 4 weeks prior to Study Day 1, or general immobility are excluded.
5. Absolute or relative contraindication to anticoagulation or treatment with apixaban, rivaroxaban, enoxaparin, or edoxaban.
6. Prior consumption of (by any route) one or more doses of aspirin (including baby aspirin), salicylate or subsalicylate, other antiplatelet drugs (e.g., ticlopidine, clopidogrel), non-steroidal anti-inflammatory drugs, fibrinolytic, or any anticoagulant within 7 days prior to Day 1 or is anticipated to require such drugs during the study.
7. Receipt of (by any route) hormonal contraception, post-menopausal hormone replacement therapy (HRT) (including over-the-counter products), or testosterone during the 4 weeks prior to Study Day 1 or is anticipated to require such drugs during the study.
8. Family history of or risk factors for a hypercoagulable or thrombotic condition, including one of the following:

   1. Factor V Leiden carrier or homozygote.
   2. Protein C, S, or ATIII activity below the normal range.
9. History of adult asthma or chronic obstructive pulmonary disease or current regular or as-needed use of inhaled medications.
10. Active HBV, HCV, or HIV-1/2 infection
11. Use of any drugs that are strong dual inhibitors or inducers of CYP3A4 and P-gp within 7 days prior to Study Day 1 or anticipated need for such drugs during the study.
12. Participation in an investigational drug study within 28 days of Day 1 or Day 1 is within 5 half-lives of the investigational compound.
13. Positive screen for drugs of abuse at Day 1 that is not explained by a prescription medication that the subject is known to be taking.
14. A medical or surgical condition that may impair drug (fXa inhibitor or andexanet) metabolism.
15. Allergy to any of the vehicle ingredients: tris, arginine, sucrose, hydrochloric acid, mannitol, and polysorbate 80.
16. Current breastfeeding or a positive pregnancy test at Screening or Day 1.
17. Any condition that could interfere with, or for which the treatment might interfere with, the conduct of the study or interpretation of the study results, or that would in the opinion of the Investigator increase the risk of the subject's participation in the study. This would include but is not limited to alcoholism, drug dependency or abuse, psychiatric disease, epilepsy, or any unexplained blackouts.
18. The subject is not judged by the study staff to have adequate bilateral venous access.
19. Unwillingness to adhere to the activity requirements of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2017-02-26 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | Day 1 through Day 7
  To evaluate the pharmacokinetics of Generation 2 process andexanet, as measured by AUC(0-∞)
Reversal | Day 1 through Day 7
  To evaluate reversal of fXa-inhibitor-mediated anticoagulation, as measured by anti-fXa activity
Safety will be evaluated by assessment of adverse events, venous thromboembolic events, physical exam findings, vital signs, oxygen saturation, fecal occult blood testing, and 12-lead ECGs. | Day 1 through Day 32
  Non-laboratory-based Endpoints
Safety will be evaluated by analyzing the following: • Hematology, chemistry & urinalysis. | Day 1 through Day 32
  Laboratory-based Endpoints
Safety will be evaluated by analyzing the following: • Antibodies to andexanet, fX, & fXa, and neutralizing antibodies | Day 1 through Day 32
  Laboratory-based Endpoints
Safety will be evaluated by analyzing the following: • TFPI, D-dimer, F1+2, thrombin-antithrombin III, and Russell's viper venom time | Day 1 through Day 32
  Laboratory-based Endpoints
Safety will be evaluated by analyzing the following: fX, fibrinogen, tissue-type plasminogen activator, plasmin-alpha2-antiplasmin complexes, thrombin activatable fibrinolysis inhibitor, beta-thromboglobulin, platelet factor 4 & soluble thrombomodulin | Day 1 through Day 32
  Laboratory-based Endpoints

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of Generation 2 process andexanet, as measured by the following PK parameter: Total area under the plasma concentration-time curve from time 0 to infinity (AUC(0 ∞) | Day 1 through Day 7
  Pharmacokinetics
Reversal | Day 1 through Day 7
  To evaluate reversal of fXa-inhibitor-mediated anticoagulation, as measured by free fraction of the fXa inhibitor
Reversal | Day 1 through Day 7
  To evaluate reversal of fXa-inhibitor-mediated anticoagulation, as measured by restoration of thrombin generation
To evaluate the pharmacokinetics of Generation 2 process andexanet, as measured by the following PK parameter: Cmax - Maximum Observed Concentration | Day 1 through Day 7
  Pharmacokinetics
To evaluate the pharmacokinetics of Generation 2 process andexanet, as measured by the following PK parameter: Tmax - Time to maximum observed plasma concentration (Tmax) | Day 1 through Day 7
  Pharmacokinetics
To evaluate pharmacokinetics of Generation 2 process andexanet as measured by following PK parameter: t1/2 - Plasma t½, determined by linear regression of the log concentration on the distribution & terminal portion of the plasma concentration-time curve | Day 1 through Day 7
  Pharmacokinetics
To evaluate the pharmacokinetics of Generation 2 process andexanet, as measured by the following PK parameter: CL - Clearance | Day 1 through Day 7
  Pharmacokinetics
To evaluate the pharmacokinetics of Generation 2 process andexanet, as measured by the following PK parameter: Vss - Volume of distribution at steady state (Vss) | Day 1 through Day 7
  Pharmacokinetics
To evaluate the pharmacokinetics of Generation 2 process andexanet, as measured by the following PK parameter: lamda z - The terminal or elimination rate constant (lamda z) | Day 1 through Day 7
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Locations (1):
- West Coast Clinical Trials, Cypress, California, United States